CLINICAL TRIAL: NCT06067685
Title: Investigating the Relationship Between Triglycerides and Fetal Overgrowth in Gestational Diabetes
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit subjects
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Gene Lee, MD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: 150494
Record Dates: First submitted 2023-09-20; First posted 2023-10-05 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Fetal Macrosomia; Obesity Complicating Childbirth; Gestational Diabetes
Keywords: fetal macrosomia; large for gestational age infant; gestational diabetes; maternal obesity; triglycerides; fatty acids; fetal overgrowth
MeSH Terms: conditions — Fetal Macrosomia; Diabetes, Gestational; Pregnancy in Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cord serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnancies with GDM and BMI > 30: Pregnancies with GDM diagnosed between 24-32 weeks and BMI > 30.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Prospective Observation only. Will record serum triglyceride, fingerstick blood triglyceride measurements, cord c-peptide, and neonatal body fat composition measurements in the first 6 months.

SUMMARY:
This is a prospective, observational study which examines the association between maternal triglycerides in the antepartum period and fetal overgrowth in pregnancies complicated by gestational diabetes. Mothers are asked to provide 2 blood samples, undergo fingerstick blood measurements, and to have their newborns measured for body fat composition in the first 6 months of life.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is a condition of impaired insulin resistance which causes increased morbidity for mothers and newborns due to fetal overgrowth. Traditionally, GDM is diagnosed with a glucose tolerance test, and treatment subsequently focuses singularly on glucose management. However, both glucose and triglycerides (TAG) are fuels for fetal overgrowth. The central hypothesis is that the most effective understanding of fetal overgrowth needs to include both carbohydrates and triglycerides. The study will focus recruitment on patients who have GDM and BMI > 35. The specific aims are 1) Determine the relationship between TAG levels during pregnancy and offspring size, 2) Explore the relationship between TAG levels during pregnancy and adipose tissue accrual (birth weight, body composition and adipose tissue distribution) from birth to six months old, and 3)Examine the relationship between maternal TAG levels and cord c-peptide levels. Mothers are asked to check their serum triglycerides at the time of diagnosis of GDM and at the end of pregnancy. Fingerstick blood measurements of triglycerides are also measured every 2 weeks at prenatal visits. At delivery, cord blood is collected. Infants are examined at 0.5, 3, and 6 months after birth.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* diagnosis of GDM between 24-32 weeks
* BMI >= 30

Exclusion Criteria:

* Conditions known to impact fetal growth.These conditions can develop after study enrollment but cannot be present at enrollment.
* autoimmune conditions treated with medication
* chronic hypertension requiring medication
* preeclampsia
* fetal growth restriction diagnosis
* smoking
* illicit drug use
* major fetal anomalies
* fetal genetic conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving prenatal care and planning to delivery at the University of Kansas Health System. Population includes significant numbers of Black and Hispanic patients. Population also includes significant numbers of self-pay and government-insured patients.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between triglyceride levels and birthweight | Newborn Day of Life 0
  Correlation coefficient

SECONDARY OUTCOMES:
Correlation coefficient between triglyceride levels and total fat mass | 0.5, 3, and 6 months
  Body fat measured by air plethysmography (PeaPod)
Correlation coefficient between triglyceride levels and body fat distribution | 0.5, 3, and 6 months
  central vs peripheral body fat measured from DEXA scan
Correlation coefficient between triglyceride levels and cord c-peptide levels | Newborn Day of Life 0
  Correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Gene T Lee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No